CLINICAL TRIAL: NCT03185026
Title: Effectiveness of the First French Psychoeducational Program for Suicidal Behavior : a Randomized Controlled Trial
Brief Title: Psychoeducation for Suicidal Behavior
Acronym: PEPSUI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: CHU Marius Lacroix, Lille, FRANCE (Unknown); CHU Gabriel Montpied, Clermont Ferrand, FRANCE (Unknown); CHU Pasteur, Nice, FRANCE (Unknown); Centre Psychothérapique de Nancy (Other); CHU Le Vinatier, Bron, FRANCE (Unknown); CHU Albert Michallon, La Tronche, FRANCE (Unknown); CHU Tarnier, Paris, FRANCE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 9808; 2017-A00571-52 (Other: Agence Nationale de Sécurité du Médicament et des produits de santé, FRANCE)
Record Dates: First submitted 2017-05-11; First posted 2017-06-14 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Suicide, Attempted; Suicidal Behavior
Keywords: Psychiatry; Suicide; Psychoeducation; Randomized controlled trial; current suicidal behavior disorder; DSM-5
MeSH Terms: conditions — Suicide, Attempted; Suicide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxation group (Active Comparator): Participants will be included in a standardized relaxation program, consisting of 10 weekly sessions lasting 2 hours. There will be 2 therapists for each patients group. Abdominal and muscular relaxation skills will be experimented.
  Interventions: Other: Relaxation group
- Psychoeducational group (Experimental): The patients will experiment the last innovating psychological skills in order to acquire the ability to engage in behaviors to manage their disease.
  Interventions: Behavioral: Interventional group : PEPSUI psychoeducational program

INTERVENTIONS:
Behavioral: Interventional group : PEPSUI psychoeducational program — The program includes 10 weekly, 2-hours sessions led by two trained animators (nurse, medical doctor/psychologist), each focusing on a specific theme or skill :
  1. Education on suicidal behavior (clinic and epidemiology), and conceptualization of the phenomenon on a matrix
  2. Education on the suicidal crisis, identification of important life areas and values for the patient, experimentation on the way to use the matrix as a decision-making tool.
  3. and 4) Self-assessment of suicidal ideations, coping strategies based on suicide ideation intensity and emotional tension (acceptation, distress tolerance, personal aid kit, and emergency care)
  5) Stress-diathesis model of suicidal behavior, innovating cognitive skills (defusion), and valued actions 6) Stress factors (psychiatric diseases and negative life events), resilience, and contact with present moment 7) Suicidal vulnerability, personal strengths 8) Social support, skills to create quality relationships
  Arms: Psychoeducational group
Other: Relaxation group — Participants will be included in a standardized relaxation program, consisting of 10 weekly sessions lasting 2 hours. There will be 2 therapists for each patients group. Abdominal and muscular relaxation skills will be experimented.
  Arms: Relaxation group

SUMMARY:
The aims of the recent World Health Organization report, highlighting that every 40 seconds a person dies from suicide somewhere in the world, are to increase awareness on the public health significance of suicide and make suicide prevention a greater priority within the global public health agenda. Across age groups, less than half of individuals at elevated suicide risk interface with some form of mental health services. Several barriers to help-seeking have been identified (maladaptive coping, lack of perceived need, beliefs about treatment effectiveness, fear of hospitalization or mistrust of providers, stigma...), which are key targets in knowledge-based interventions on suicide. Psychoeducational programs have shown effectiveness in prevention relapse for several mental disorders such as schizophrenia, bipolar disorder or recurrent depressive disorder, improving treatment adherence and self-confidence in coping with symptoms of the disease. They are highly recommended for addressing adherence problems in patients with serious and persistent mental illness. Only one team has published a study protocol for a controlled trial assessing a 10 group sessions psychoeducational program for prevention in patients having a suicide history, in a one-year follow-up. Interestingly, diagnosis-mixed group psychoeducation have shown superiority than an unspecific intervention add-on routine care, on the suicide prevention and compliance for severe psychiatric disorders. Those psychoeducational-specific elements are namely the interactive transfer of illness and treatment-related knowledge and management/coping - cognitive/behavioral - strategies, as defined by the National Institute for Health and Care Excellence)-Guidelines (NICE). Notably, as several psychiatric diagnoses are associated with suicidal behavior (SB), coping strategies have to target processes that overlap among these psychiatric disease, as well as suicidal vulnerability. Acceptance and Commitment Therapy (ACT), a "third wave" behavioral therapy, targets experiential avoidance and psychological flexibility, at the core of psychiatric disorders. Interestingly, in patients with a history of suicidal depression, training in mindfulness can help to weaken suicidal thinking associated with depressive symptoms , and thus reduce an important vulnerability for relapse to suicidal depression. ACT would also increase intrinsic motivation for daily life action (i.e. reasons for living and acting). Then, the functional analysis (matrix) used in ACT seems to be an useful tool to help patient in decision making, a neuropsychological factor impaired in suicidal patients. Finally, acceptance and commitment group therapy has suggested effectiveness in reducing intensity and frequency of suicidal thoughts, through improvement in acceptance, in high risk suicidal patients. As compared with ACT, Dialectical behavior therapy (DBT) teaches added distress tolerance in view of survive the crisis. DBT is the most validated therapy for borderline personality disorder, the mental disorder the most associated with SB . Notably, group skills training is the most effective component in DBT for preventing suicidal behavior in borderline patients with high suicidal risk. Furthermore, interventions based on positive psychology have suggested efficacy in reducing depressive symptoms and suicidal ideation. Notably, in a recent pilot study, positive psychology exercises delivered to suicidal inpatients were feasible and associated with short-term gains improvement in optimism and hopelessness. Finally, as altered social link and sense of belonging have been widely involved in SB, relationship skills are an interesting positive psychology area for suicide prevention program.

Psychoeducational program integrating knowledge as well the last innovating cognitive-behavioral coping strategies for SB is of major interest in suicide prevention.

Investigators developed the first French program of suicide psychoeducation called "PEPSUI". The aim of this innovating program is to teach patients the more recent knowledge about suicidal behaviour (SB) and effective treatments, through didactic and interactive sessions. Thus, the objective is to conduct the patients to become experts and actors of their disease, increasing adherence to treatment. Besides, the patients will experiment the last innovating psychological skills to cope with unpleasant emotions and thoughts (including suicidal thoughts), distress tolerance skills and crisis strategies, and identify personal purpose in life and learn positive psychological skills in order to anchor with meaningful and pleasant components in life. Thus, this program will include skills from ACT, DBT and positive psychology. Finally, this primary care research is about a program which aim at improving accessibility to mental health services, care adherence and continuity for suicidal patients.

DETAILED DESCRIPTION:
The project aims at to compare the effectiveness on suicide re-attempt rate reduction at 2-years follow-up of add-on PEPSUI psychoeducational program versus relaxation program in patients having attempted suicide in the past year

Secondary, the project aims to compare between add-on psychoeducational program and relaxation:

* Interrupted or aborted suicide attempt rate reduction during the follow-up
* Severity and intensity of suicide ideation: at post-treatment, and at 6, 12, 18 and 24 months after the intervention (and the evolution between pre and each post-intervention point)
* Intensity of suicidal intent: at post-treatment, and at 6, 12, 18 and 24 months after the intervention (and the evolution between pre and each post-intervention point)
* Adherence to treatment and perceived utility of mental health services: at post-treatment, and at 6, 12, 18 and 24 months after the intervention (and the evolution between pre and each post-intervention point)
* Levels of depression, anxiety, psychological pain and hopelessness: at post-treatment, and at 6, 12, 18 and 24 months after the intervention (and the evolution between pre and each post-intervention point)
* Global functioning and quality of life: at post-treatment, and at 6, 12, 18 and 24 months after the intervention (and the evolution between pre and each post-intervention point)
* Subjective social support: at post-treatment, and at 6, 12, 18 and 24 months after the intervention (and the evolution between pre and each post-intervention point)
* The need to emergency psychiatric consultation and psychiatric hospitalisation for suicidal ideation: at post-treatment, and at 6, 12, 18 and 24 months after the intervention (and the evolution between pre and each post-intervention point)
* Acceptance, contact with present moment and meaning in life: at post-treatment, and at 6, 12, 18 and 24 months after the intervention (and the evolution between pre and each post-intervention point)
* Satisfaction and adherence to the intervention: at post-treatment (likert scale).

  500 patients suffering from current suicidal behavior disorder (according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) will be recruited, i.e. having attempted to suicide in the past year. Eligible patients will be randomized in one of the two arms: add-on psychoeducation or add-on relaxation (computer-generated randomisation in a 1 :1 ratio).

Sociodemographic data, psychiatric diagnoses using Mini-International Neuropsychiatric Interview (M.I.N.I.) and pharmacological treatment will be also recorded.

An independent researcher not involved in the study will perform the allocation. Each patient will be evaluated at baseline (pre intervention V1) and followed-up during 24 months after treatment completion, with 5 visits: post intervention (V2) 6 months (V3), 12 months (V4), 18 months (V5) and 24 months (V6) after the intervention. Blind trained evaluators will assess patients. Patients will be told to avoid saying their group of allocation to the evaluator.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years
* Having a current suicidal behaviour disorder according to DSM-5 (APA, 2013), i.e. history of suicidal attempt in the past year
* Able to speak, read and understand French.
* Able to give written informed consent
* Having signed informed consent
* Must belong to social safety system

Exclusion Criteria:

* Having a current or past diagnosis of an organic mental disorder
* Having a lifetime history of schizophrenia
* Having a mental retardation
* Planned longer stay outside the region that prevents compliance with the visit plan
* Deprived of liberty Subject (by judicial or administrative decision)
* Protected by law (guardianship)
* Current exclusion period in relation to another protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-09-06 (Actual); Primary Completion 2026-05-06 (Estimated); Study Completion 2026-05-06 (Estimated)

PRIMARY OUTCOMES:
Suicide re-attempt rate reduction using the Columbia Suicide Severity Rating Scale (C-SSRS) | At 2 years after the intervention
  Comparison of suicide re-attempt rate reduction, at 2 years follow-up, between PEPSUI and relaxation groups.

SECONDARY OUTCOMES:
Interrupted suicide attempt rate reduction using the C-SSRS | At 2 years after the intervention
  Comparison of suicide re-attempt rate reduction, at 2 years follow-up, between PEPSUI and relaxation groups.
Aborted suicide attempt rate reduction using the C-SSRS | At 2 years after the intervention
  Comparison of suicide re-attempt rate reduction, at 2 years follow-up, between PEPSUI and relaxation groups.
Severity of suicide ideation using the C-SSRS | At one week after the intervention
  Comparison of the severity of suicide ideation between pre-intervention and post-intervention (one week after the last session of the intervention) within the two groups (PEPSUI versus Relaxation).
Severity of suicide ideation using the C-SSRS | At 6 months after the intervention
  Comparison of the severity of suicide ideation between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation)
Severity of suicide ideation using the C-SSRS | At 12 months after the intervention
  Comparison of the severity of suicide ideation between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
Severity of suicide ideation using the C-SSRS | At 18 months after the intervention
  : Comparison of the severity of suicide ideation between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
Severity of suicide ideation using the C-SSRS | At 24 months after the intervention
  Comparison of the severity of suicide ideation between pre-treatment and 24 months post-intervention within the two groups (PEPSUI vs Relaxation).
Severity of suicide ideation evaluated by the likert scales from 0 (none) to 10 (maximum possible suicidal ideation) | At one week after the intervention
  Comparison of the severity of suicide ideation between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
Severity of suicide ideation evaluated by the likert scales from 0 (none) to 10 (maximum possible suicidal ideation) | At 6 months after the intervention
  Comparison of the severity of suicide ideation between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
Severity of suicide ideation evaluated by the likert scales from 0 (none) to 10 (maximum possible suicidal ideation) | At 12 months after the intervention
  Comparison of the severity of suicide ideation between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
Severity of suicide ideation evaluated by the likert scales from 0 (none) to 10 (maximum possible suicidal ideation) | At 18 months after the intervention
  Comparison of the severity of suicide ideation between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
Severity of suicide ideation evaluated by the likert scales from 0 (none) to 10 (maximum possible suicidal ideation) | At 24 months after the intervention
  Comparison of the severity of suicide ideation between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
Intensity of suicide ideation using the Columbia-Suicide Severity Rating Scale (C-SSRS) | At one week after the intervention
  Comparison of the intensity of suicide ideation between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
Intensity of suicide ideation using the Columbia-Suicide Severity Rating Scale (C-SSRS) | At 6 months after the intervention
  Comparison of the intensity of suicide ideation between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
Intensity of suicide ideation using the Columbia-Suicide Severity Rating Scale (C-SSRS) | At 12 months after the intervention
  Comparison of the intensity of suicide ideation between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
Intensity of suicide ideation using the Columbia-Suicide Severity Rating Scale (C-SSRS) | At 18 months after the intervention
  Comparison of the intensity of suicide ideation between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
Intensity of suicide ideation using the Columbia-Suicide Severity Rating Scale (C-SSRS) | At 24 months after the intervention
  Comparison of the intensity of suicide ideation between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
Intensity of suicide ideation using the likert scales, from 0 (none) to 10 (maximum possible suicidal ideation) | At one week after the intervention
  Comparison of the intensity of suicidal intent between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
Intensity of suicide ideation using the likert scales, from 0 (none) to 10 (maximum possible suicidal ideation) | At 6 months after the intervention
  Comparison of the intensity of suicidal intent between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
Intensity of suicide ideation using the likert scales, from 0 (none) to 10 (maximum possible suicidal ideation) | At 12 months after the intervention
  Comparison of the intensity of suicidal intent between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
Intensity of suicide ideation using the likert scales, from 0 (none) to 10 (maximum possible suicidal ideation) | At 18 months after the intervention
  Comparison of the intensity of suicidal intent between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
Intensity of suicide ideation using the likert scales, from 0 (none) to 10 (maximum possible suicidal ideation) | At 24 months after the intervention
  Comparison of the intensity of suicidal intent between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
Adherence to treatment using the Medication Adherence Rating Scale (MARS) | At one week after the intervention
  Comparison of the pharmacological adherence between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
Adherence to treatment using the Medication Adherence Rating Scale (MARS) | At 6 months after the intervention
  Comparison of the pharmacological adherence between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
Adherence to treatment using the Medication Adherence Rating Scale (MARS) | At 12 months after the intervention
  Comparison of the pharmalogical adherence between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
Adherence to treatment using the Medication Adherence Rating Scale (MARS) | At 18 months after the intervention
  Comparison of the pharmacological adherence between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation)
Adherence to treatment using the Medication Adherence Rating Scale (MARS) | At 24 months after the intervention
  Comparison of the pharmacological adherence between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
Perceived utility of mental health services using the likert scales rating from 0 (not useful at all) to 10 (very useful) | At one week after the intervention
  Comparison of the number of missed consultations between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
Perceived utility of mental health services using the likert scales rating from 0 (not useful at all) to 10 (very useful) | At 6 months after the intervention
  Comparison of the number of missed consultations between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
Perceived utility of mental health services using the likert scales rating from 0 (not useful at all) to 10 (very useful) | At 12 months after the intervention
  Comparison of the number of missed consultations between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
Perceived utility of mental health services using the likert scales rating from 0 (not useful at all) to 10 (very useful) | At 18 months after the intervention
  Comparison of the number of missed consultations between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
Perceived utility of mental health services using the likert scales rating from 0 (not useful at all) to 10 (very useful) | At 24 months after the intervention
  Comparison of the number of missed consultations between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
Depression intensity using the Inventory of Depressive Symptomatology (IDS-C30) | At one week after the intervention
  Comparison of the intensity of depression between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
Depression intensity using the Inventory of Depressive Symptomatology (IDS-C30) | At 6 months after the intervention
  Comparison of the intensity of depression between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
Depression intensity using the Inventory of Depressive Symptomatology (IDS-C30) | At 12 months after the intervention
  Comparison of the intensity of depression between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
Depression intensity using the Inventory of Depressive Symptomatology (IDS-C30) | At 18 months after the intervention
  Comparison of the intensity of depression between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
Depression intensity using the Inventory of Depressive Symptomatology (IDS-C30) | At 24 months after the intervention
  Comparison of the intensity of depression between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
Anxiety state using the State-Trait Anxiety Inventory (STAI-State) | At one week after the intervention
  Comparison of the state of anxiety between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
Anxiety state using the State-Trait Anxiety Inventory (STAI-State) | At 6 months after the intervention
  Comparison of the state of anxiety between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
Anxiety state using the State-Trait Anxiety Inventory (STAI-State) | At 12 months after the intervention
  Comparison of the state of anxiety between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
Anxiety state using the State-Trait Anxiety Inventory (STAI-State) | At 18 months after the intervention
  Comparison of the state of anxiety between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
Anxiety state using the State-Trait Anxiety Inventory (STAI-State) | At 24 months after the intervention
  Comparison of the state of anxiety between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
Psychological pain using the Likert scales from 0 (none) to 10 (maximum possible pain) | At one week after the intervention
  Comparison of the psychological pain between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
Psychological pain using the Likert scales from 0 (none) to 10 (maximum possible pain) | At 6 months after the intervention
  Comparison of the psychological pain between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
Psychological pain using the Likert scales from 0 (none) to 10 (maximum possible pain) | At 12 months after the intervention
  Comparison of the psychological pain between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
Psychological pain using the Likert scales from 0 (none) to 10 (maximum possible pain) | At 18 months after the intervention
  Comparison of the psychological pain between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
Psychological pain using the Likert scales from 0 (none) to 10 (maximum possible pain) | At 24 months after the intervention
  Comparison of the psychological pain between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
Hopelessness using the Beck Hopelessness Scale (BHS) | At one week after the intervention
  Comparison of the hopelessness between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
Hopelessness using the Beck Hopelessness Scale (BHS) | At 6 months after the intervention
  Comparison of the hopelessness between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
Hopelessness using the Beck Hopelessness Scale (BHS) | At 12 months after the intervention
  Comparison of the hopelessness between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
Hopelessness using the Beck Hopelessness Scale (BHS) | At 18 months after the intervention
  Comparison of the hopelessness between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
Hopelessness using the Beck Hopelessness Scale (BHS) | At 24 months after the intervention
  Comparison of the hopelessness between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
Global functioning using the Functioning Assessment Short Test (FAST) | At one week after the intervention
  Comparison of the global functioning between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
Global functioning using the Functioning Assessment Short Test (FAST) | At 6 months after the intervention
  Comparison of the global functioning between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
Global functioning using the Functioning Assessment Short Test (FAST) | At 12 months after the intervention
  Comparison of the global functioning between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
Global functioning using the Functioning Assessment Short Test (FAST) | At 18 months after the intervention
  Comparison of the global functioning between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
Global functioning using the Functioning Assessment Short Test (FAST) | At 24 months after the intervention
  Comparison of the global functioning between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
Quality of life evaluated by the World Health Organization Quality Of Life measure (WHOQOL-BREF) instrument | At one week after the intervention
  Comparison of the quality of life between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
Quality of life evaluated by the World Health Organization Quality Of Life measure (WHOQOL-BREF) instrument | At 6 months after the intervention
  Comparison of the quality of life between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
Quality of life evaluated by the World Health Organization Quality Of Life measure (WHOQOL-BREF) instrument | At 12 months after the intervention
  Comparison of the quality of life between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
Quality of life evaluated by the World Health Organization Quality Of Life measure (WHOQOL-BREF) instrument | At 18 months after the intervention
  Comparison of the quality of life between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
Quality of life evaluated by the World Health Organization Quality Of Life measure (WHOQOL-BREF) instrument | At 24 months after the intervention
  Comparison of the quality of life between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
Subjective social support using a Likert scale, from 0 (very poor quality) to 10 (excellent quality) | At one week after the intervention
  Comparison of the subjective social support between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
Subjective social support using a Likert scale, from 0 (very poor quality) to 10 (excellent quality) | At 6 months after the intervention
  Comparison of the subjective social support between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
Subjective social support using a Likert scale, from 0 (very poor quality) to 10 (excellent quality) | At 12 months after the intervention
  Comparison of the subjective social support between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
Subjective social support using a Likert scale, from 0 (very poor quality) to 10 (excellent quality) | At 18 months after the intervention
  Comparison of the subjective social support between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
Subjective social support using a Likert scale, from 0 (very poor quality) to 10 (excellent quality) | At 24 months after the intervention
  Comparison of the subjective social support between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
The need to emergency psychiatric consultation for suicidal ideation | At one week after the intervention
  Comparison of need to emergency psychiatric consultation between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
The need to emergency psychiatric hospitalisation for suicidal ideation | At one week after the intervention
  Comparison of need to emergency psychiatric hospitalisation between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
The need to emergency psychiatric consultation for suicidal ideation | At 6 months after the intervention
  Comparison of need to emergency psychiatric consultation between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
The need to emergency psychiatric hospitalisation for suicidal ideation | At 6 months after the intervention
  Comparison of need to emergency psychiatric hospitalisation between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
The need to emergency psychiatric consultation for suicidal ideation | At 12 months after the intervention
  Comparison of need to emergency psychiatric consultation between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
The need to emergency psychiatric hospitalisation for suicidal ideation | At 12 months after the intervention
  Comparison of need to emergency psychiatric hospitalisation between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
The need to emergency psychiatric consultation for suicidal ideation | At 18 months after the intervention
  Comparison of need to emergency psychiatric consultation between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
The need to emergency psychiatric hospitalisation for suicidal ideation | At 18 months after the intervention
  Comparison of need to emergency psychiatric hospitalisation between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
The need to emergency psychiatric consultation for suicidal ideation | At 24 months after the intervention
  Comparison of need to emergency psychiatric consultation between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
The need to emergency psychiatric hospitalisation for suicidal ideation | At 24 months after the intervention
  Comparison of need to emergency psychiatric hospitalisation between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
Acceptance assessment using the acceptance and Action Questionnaire (AAQII) | At one week after the intervention
  Comparison of the acceptance between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
Acceptance assessment using the acceptance and Action Questionnaire (AAQII) | At 6 months after the intervention
  Comparison of the acceptance between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
Acceptance assessment using the acceptance and Action Questionnaire (AAQII) | At 12 months after the intervention
  Comparison of the acceptance between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
Acceptance assessment using the acceptance and Action Questionnaire (AAQII) | At 18 months after the intervention
  Comparison of the acceptance between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
Acceptance assessment using the acceptance and Action Questionnaire (AAQII) | At 24 months after the intervention
  Comparison of the acceptance between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
Contact with the present moment assessment using the Mindful Attention Awareness Scale (MAAS) | At one week after the intervention
  Comparison of the contact with the present moment between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
Contact with the present moment assessment using the Mindful Attention Awareness Scale (MAAS) | At 6 months after the intervention
  Comparison of the contact with the present moment between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
Contact with the present moment assessment using the Mindful Attention Awareness Scale (MAAS) | At 12 months after the intervention
  Comparison of the contact with the present moment between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
Contact with the present moment assessment using the Mindful Attention Awareness Scale (MAAS) | At 18 months after the intervention
  Comparison of the contact with the present moment between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
Contact with the present moment assessment using the Mindful Attention Awareness Scale (MAAS) | At 24 months after the intervention
  Comparison of the contact with the present moment between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
Meaning in life assessment using the Life Regard Index: (LRI) | At one week after the intervention
  Comparison of the meaning in life between pre-treatment and one week post-intervention within the two groups (PEPSUI versus Relaxation).
Meaning in life assessment using the Life Regard Index: (LRI) | At 6 months after the intervention
  Comparison of the meaning in life between pre-treatment and 6 months post-intervention within the two groups (PEPSUI versus Relaxation).
Meaning in life assessment using the Life Regard Index: (LRI) | At 12 months after the intervention
  Comparison of the meaning in life between pre-treatment and 12 months post-intervention within the two groups (PEPSUI versus Relaxation).
Meaning in life assessment using the Life Regard Index: (LRI) | At 18 months after the intervention
  Comparison of the meaning in life between pre-treatment and 18 months post-intervention within the two groups (PEPSUI versus Relaxation).
Meaning in life assessment using the Life Regard Index: (LRI) | At 24 months after the intervention
  Comparison of the meaning in life between pre-treatment and 24 months post-intervention within the two groups (PEPSUI versus Relaxation).
Satisfaction of the intervention using the Likert scales rating from 0 (not useful at all) to 10 (very useful) | One week after last session of the intervention within 15 days.
  Evaluation of the satisfaction about the intervention within the two groups (PEPSUI versus Relaxation).
Adherence to the intervention (psychoeducational and relaxation ): number of sessions performed by the patient | At one week after the intervention
  Comparison of adherence to the intervention within the two groups (PEPSUI versus Relaxation) assessed by the number of sessions performed by patients

CONTACTS AND LOCATIONS:
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793